CLINICAL TRIAL: NCT04252482
Title: Validation of Sleep Healthcare System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201802034RIPD
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: basal metabolism; body weight; energy intake; energy metabolism; insulin resistance
MeSH Terms: conditions — Sleep Apnea, Obstructive; Body Weight; Insulin Resistance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Use of CPAP device (Experimental): CPAP 12 weeks
  Interventions: Device: CPAP
- Usual care (No Intervention): Usual care 12 weeks

INTERVENTIONS:
Device: CPAP — Auto-CPAP treatment (AirSense™ 10 Autoset™, ResMed Inc., Australia) for 12 weeks
  Arms: Use of CPAP device

SUMMARY:
The present project aims to that examine the interplay between sleep duration circadian phase, and metabolic regulation. The impact of CPAP therapy on metabolic regulation is assessed with a RCT. Patients were enrolled form referral to sleep clinic for suspect obstructive sleep apnea (OSA). Subjects with hypopnea index (AHI) >=15/h are randomly allocated to the usual care or Auto-PAP (APAP) therapy then reevaluated after 12th week. The CPAP effect are measured with the comparison of changes in outcomes between usual care and APAP therapy.

DETAILED DESCRIPTION:
Enrolled participants undertake pre-randomization evaluations. That included standard questionnaire, eating behavior, International Physical Activity Questionnaire (IPAQ)-short form, 3-day dietary intake, and 7-day sleep log, 24-hr ambulatory blood pressure, and 7-day Actiwatch. Within one week after completion, participants underwent repeated polysomnography (PSG) to confirm the diagnosis of OSA. The basal metabolic rate (BMR) and body composition (BC), and blood sampling are conducted in the morning next to overnight PSG and BMR.

Once the pre-randomization evaluation was completed and the AHI >=15/h was confirmed, participants are randomly allocated to the usual care or auto-CPAP treatment (AirSense™ 10 Autoset™, ResMed Inc., Australia) for 12 weeks. Participants had two follow-up visits at 4th and 12th week and were reevaluated with the same measurements as pre-randomization Enrolled participants are randomized into CPAP or usual care. The randomization is generated by the staff of the Department of Biostatistics independent of subject enrolment. A block-randomized assignment with a block size of four is used. Consecutive patients are assigned to the allocation according to the randomization schedule by the study nurse. Investigators who assess outcome are blinded to the allocation assignment. Preset-dropout criteria: Defaulting clinic visits at 4th and 12-week, re-assessment, and clinical exacerbations requiring medical attention.

Participants starting CPAP are instructed to use the device for >=6hr/night. PAP compliance is assessed as the average usage hours per night which is objectively recorded on the devices with a built-in compliance meter. Compliance data are downloaded by medical staff at every clinic visit. The good compliance is defined as usage>= 4hr/night in 70% days of total period.

ELIGIBILITY:
Inclusion Criteria:

1. >=20 year-old
2. patients with moderate-severe OSA (AHI≥15/hr)

Exclusion Criteria:

1. skin allergy
2. wrist tattoos
3. BMI≧40 kg/m2
4. Neurological Disorders(Infection, Stroke, ALS, Myopathy, Brain tumor and Encephalitis)
5. Internal Diseases(cardiovascular disease or coronary artery disease was poorly controlled
6. chronic heart failure(including NYHA class 3 or more than NYHA class 3)
7. COPD(FEV1/FVC<70)
8. Hyperthyroidism or Hypothyroidism
9. Primary Aldosteronism
10. Chronic Kidney Disease(eGFR<30)
11. Acromegaly and Parkinson's disease)
12. Psychosis(Schizophrenia, bipolar disorder and depression)
13. Autoimmune disease(System Lupus Erythematosus, Rheumatoid arthritis, Sarcoidosis, Crohn's disease and Ulcerative Colitis)
14. Cancer(in last 5 years)
15. Have been diagnosed with obstructive sleep apnea
16. other sleep disorder(Narcolepsy, insomnia and RBD)
17. Use anti-inflammatory drugs(in last 2 weeks)
18. Illiterate
19. shift worker
20. has been Spinal Surgery and move difficult
21. professional driver has severe drowsiness

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
The difference before and after the treatment of BMR (REE) | 12 weeks
  The difference in BMR(Basal metabolic rate) between the CPAP group and the usual care group. The comparison item is REE(Resting Energy Expenditure) (kcal/day)

SECONDARY OUTCOMES:
The difference before and after the treatment of BC(total fat mass and fat free mass) | 12 weeks
  Compare the total fat mass and fat free mass between the usual care group and the CPAP group to demonstrate the effectiveness before and after treatment. The units for total fat mass and fat free mass are both in kg.
The difference before and after the treatment of energy intake and percentage of nutrients | 12 weeks
  The difference before and after treatment is represented by comparing the calorie intake from the three-day food diaries between the usual care group and the CPAP group. The evaluation unit is total calories (% nutrition).
The difference before and after the treatment of eating behavior | 12 weeks
  Compare the eating behavior between the usual care group and the CPAP group to demonstrate the differences before and after treatment. Eating behavior includes cognitive restraint, uncontrolled eating, and emotional eating, which are assessed using the 18 items of the Three-Factor Eating Questionnaire(TFEQ).
The difference before and after the treatment of 24h blood pressure | 12 weeks
  The difference in 24-h systolic, diastolic(mmHg), and mean BP(mmHg) between the CPAP group and the usual care group.
The difference before and after the treatment of sleep parameters | 12 weeks
  The difference before and after treatment is represented by comparing sleep parameters (hours of sleep, TIB, sleep efficiency) between the usual care group and the CPAP group. The activity levels are measured using an Actiwatch (Spectrum Plus, Philips Respironics, USA).
The difference before and after the treatment of Physical Activity(PA) | 12 weeks
  Compare the difference between participants' self-reported International Physical Activity Questionnaire-Short Form(IPAQ-SF) questionnaire and the objectively measured physical activity from the Actiwatch to demonstrate the effectiveness of CPAP treatment. The IPAQ-SF primarily analyzes total physical activity (MET time/week) and the percentage of vigorous-intensity activity, while the Actiwatch analyzes the average activity count per minute measured by the device.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Lin Lee, M.D., PhD, Principal Investigator — Department of Internal Medicine
Locations (1):
- Center of sleep disorders, National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee PL, Chien MY, Lai SR, Gooley JJ, Feng HC, Chen SK, Lin MT, Chen YH, Chiu HC, Liu PK, Ku BW, Wang SM, Chang CH, Yang WS, Yu CJ. Continuous positive airway pressure effects on energy expenditure, intake, hormonal regulation, and body composition: a randomized trial. Sleep. 2026 Jan 13;49(1):zsaf259. doi: 10.1093/sleep/zsaf259. PMID 40874641
- [Derived] Liu PK, Ting N, Chiu HC, Lin YC, Liu YT, Ku BW, Lee PL. Validation of photoplethysmography- and acceleration-based sleep staging in a community sample: comparison with polysomnography and Actiwatch. J Clin Sleep Med. 2023 Oct 1;19(10):1797-1810. doi: 10.5664/jcsm.10690. PMID 37338335